CLINICAL TRIAL: NCT07092904
Title: iTide 2 - STEMI Follow-up Study
Brief Title: Myocardial Infarction Safe Emergency Medicine Accompanying Study: Providing Reperfusion Therapy Within the Recommended Time Limits
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 904338
Record Dates: First submitted 2025-04-08; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Infarction
Keywords: Acute myocardial infarction; Pharmacoinvasive; Reperfusion therapy; Emergency medicine; Prehospital thrombolysis; primary PCI
MeSH Terms: conditions — Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with acute ST elevation myocardial infarction in our region, all-comers: The patients are not subjected to any intervention for the study purpose.

SUMMARY:
The project is a prospective observational study with the aim of system improvement. It represents accompanying research in connection with the implementation of Safe Emergency Medicine , - an initiative under the auspices of the board of The North Norway Regional Health Authority and The Municipal Health Consortium that aims to provide faster and better treatment to patients with common, serious and time-critical conditions.

The focus of the study is the decision-making process and implementation of treatment algorithms for all patients with acute ST-elevation myocardial infarction (STEMI) in the regional health trust's admission area. The data sources are 1) structured telephone interviews with providers and decision-makers and 2) electronic medical records (AMIS, DIPS, prehospital medical records from emergency departments, ambulance medical records). The analyses will form the basis for recommendations for improvements in procedures, training and organization.

DETAILED DESCRIPTION:
STEMI Follow-up Study. Project Plan

Project manager Senior consultant prof. Kristian Bartnes, The Division of Cardiothoracic and Pulmonary Medicine, the University Hospital North Norway (UNN) and UiT The Arctic University of Norway

Team members Senior consultant prof. Mads Gilbert, The Division of Emergency Medicine, UNN and UiT The Arctic University of Norway Senior consultant Jan Mannsverk, Department of Cardiology, UNN Student of medicine Maryam Amri, UNN and UiT The Arctic University of Norway Project manager Safe Emergency Medicine Stein-G. Widding, UNN

Project summary The project is a prospective observational study with the aim of system improvement. It represents accompanying research in connection with the implementation of Safe Emergency Medicine , - an initiative under the auspices of the board of The North Norway Regional Health Authority and The Municipal Health Consortium that aims to provide faster and better treatment to patients with common, serious and time-critical conditions.

The study focuses on the decision-making process and implementation of treatment algorithms for all patients with acute ST-elevation myocardial infarction (STEMI) in the regional health trust's admission area. The data sources are 1) structured telephone interviews with providers and decision-makers and 2) electronic medical records (AMIS, DIPS, prehospital medical records from emergency departments, ambulance medical records). The analyses will form the basis for recommendations for improvements in procedures, training and organization.

Purpose The primary goal is to improve emergency care so that more patients survive STEMI with preserved cardiac function.

Quality improvement < 50% of STEMI patients in Northern Norway receive reperfusion treatment (thrombolysis or primary PCI) within the recommended time intervals (2023: Northern Norway 45%, the country as a whole 69%) . Previous studies and registry data3 have identified several targets for improvement efforts: i) more efficient on-site workflow, ii) faster and more precise communication among the emergency care providers, iii) more efficient decision-making, iv) competence enhancement.

Patient safety Loss of time leads to loss of myocardium and in some cases death, or survival with chronic heart failure.

Generalization value Improving quality for one patient category will also benefit other categories within the same treatment system. And extensive, resource-intensive initiatives should be evaluated and adjusted accordingly.

Safe emergency medicine aims to provide faster and better treatment of patients with common, serious emergency medical conditions (heart attack, stroke, sepsis) with. The initiative is backed by the board of The Regional Health Trust and The Municipal Health Consortium and is being gradually implemented throughout the region. The current project is an accompanying research-initiative aimed at one of the relevant patient categories. Other categories with time-critical conditions will benefit from the experiences we gain from the STEMI segment, since they depend on the same system.

Material/method Inclusion All patients with a diagnosis of acute STEMI in the catchment area of The North Norway Regional Health Authority's hospitals in the period approx. May 1st - October 31st 2025.

Privacy and ethics The protocol is submitted to the hospital's data protection officer and the Regional Ethics Committee for approval.

Parameters Patient data Clinical course for 1 month from onset, with exact time intervals and description of interventions and treatment results. Data are collected from electronic sources (AMIS, emergency room physician's notes, ambulance records, air ambulance records, DIPS, MetaVision, diagnostic imaging systems).

Decision-making process For all patients, the agencies involved in communication and decisions about treatment modality and location are described, from the first contact with the health service until the start of reperfusion therapy (or decision to forgo it). Effective and consistent use of multi-party conversation has been identified as a critical vulnerability and will be given special emphasis in the analysis.

Time spent, form of communication (emergency network radio, telephone, multi-party call or sequential, etc.) are recorded.

Data are collected through structured telephone interviews with therapists and decision-makers within 2 days of patient inclusion, based on a self-developed template.

Analyses Statistical analyses of categorical and continuous variables are performed using electronic tools (SPSS, Excel), including time-to-event and regression analyses.

Statistical strength A 40% improvement for the primary endpoint from 2021 to 2025 would be significant at the 5% level.

Primary endpoint Proportion of STEMI patients who receive reperfusion therapy within the recommended time.

Secondary endpoints Extent of aim achievement (proportion of patients within the recommended time interval) for process indicators in the acute course of STEMI: time from first medical contact to i) ECG recording, ii) STEMI diagnosis, iii) treatment decision.

Degree of compliance with time intervals described in Safe Emergency Medicine and guidelines for prehospital communication.

Dissemination/publication of results The results will be published in a scientific journal and used in a master's thesis for medical student(s), shared at professional meetings and included in improvement work within the framework of the regional Safe Acute Medicine project.

ELIGIBILITY:
Inclusion Criteria:

* Patient with the diagnosis of acute ST elevation myocardial infarction located within the uptake area of the Northern Norway Regional Health Authority

Exclusion Criteria:

* Patient declines use of data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute ST elevation myocardial infarction within the municipalities of Nordland, Troms and Finnmark.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with acute ST elevation myocardial infarction who receive reperfusion therapy within the recommended time intervals. | Inclusion will be performed during 6 months from September 1st 2025 - March 1st 2026. Each patient will be monitored for 1 month after enrollment (baseline). The interval from the diagnostic ECG recording to reperfusion therapy initiation is reported.
  Internationally approved guidelines provide clear, evidence-based time interval recommendations for receiveing rapid reperfusion therapy, either by fibrinolytic medication or primary percutaneous coronary intervention. The primary endpoint adresses the extent of aim fulfillment.

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Bartnes, PhD, Principal Investigator — University hospital North Norway; Mads F Gilbert, PhD, Study Chair — University hospital North Norway
Locations (1):
- University hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uleberg B, Bonaa KH, Govatsmark RES, Olsen F, Jacobsen BK, Stensland E, Hauglann B, Vonen B, Forde OH. Exploring variation in timely reperfusion treatment in ST-segment elevation myocardial infarction in Norway: a national register-based cohort study. BMJ Open. 2024 Feb 17;14(2):e081301. doi: 10.1136/bmjopen-2023-081301. PMID 38367969
- [Background] The Norwegian Registry for Myocardial Infarction. Annual Report for 2023. https://www.kvalitetsregistre.no/sites/default/files/2024-06/Årsrapport%202023_Norsk%20hjert
- [Background] Hansen, AS (2021). Treatment and outcome for patients with ST-elevation myocardial infarction in Norway. Are there differences in the management and outcome of STEMI within Norway and compared to other Nordic countries? (Master's thesis, UiT Arctic University of Norway)
- [Background] Bartnes K, Albrigtsen H, Iversen JM, Brovold H, Moller NH, Wembstad B, Arstad F, Kristensen AH, Cortis J, Olsen SJ, Nygaard SNS, Kindler SG, Moe O, Hansen C, Mannsverk JT. The Barriers to Rapid Reperfusion in Acute ST-Elevation Myocardial Infarction. Cardiol Ther. 2022 Dec;11(4):559-574. doi: 10.1007/s40119-022-00281-7. Epub 2022 Oct 6. PMID 36203049
- [Background] Mannsverk J, Steigen T, Wang H, Tande PM, Dahle BM, Nedrejord ML, Hokland IO, Gilbert M. Trends in clinical outcomes and survival following prehospital thrombolytic therapy given by ambulance clinicians for ST-elevation myocardial infarction in rural sub-arctic Norway. Eur Heart J Acute Cardiovasc Care. 2019 Feb;8(1):8-14. doi: 10.1177/2048872617748550. Epub 2017 Dec 19. PMID 29256635